CLINICAL TRIAL: NCT00836836
Title: Evaluation Of The Efficacy Of The Modified Atkins Diet In Children With Refractory Epilepsy: A Randomized Controlled Trial.
Brief Title: Modified Atkins Diet in Childhood Epilepsy
Acronym: mAD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: Council of Scientific and Industrial Research, India (Other Government)
Responsible Party: Principal Investigator, Suvasini Sharma, Senior Research Associate, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ModAtkins
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Refractory Childhood Epilepsy
Keywords: Childhood epilepsy; ketogenic diet
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Modified Atkins diet arm-In this arm, the children will start the modified Atkins diet after a 4-week baseline period, during which daily seizure log will be maintained. Anti-epileptic medications will remain unchanged during the 3 month trial period, unless the change in AED regimen is medically indicated; e.g. drug side effects or status epilepticus; in which case standard therapy will be provided.
  Interventions: Other: Modified Atkins diet
- 2 (No Intervention): No Intervention arm- After the 4-week baseline period, this group will receive their normal diet with no dietetic input, and remain on the same on-going antiepileptic medication for the 3 months. Anti-epileptic medications will remain unchanged during the 3 month trial period, unless the change in AED regimen is medically indicated; e.g. drug side effects or status epilepticus; in which case standard therapy will be provided.
  At the end of three months, patients in this arm will be offered the option of the modified Atkins diet treatment.
  This group will not receive any dietetic input

INTERVENTIONS:
Other: Modified Atkins diet — Modified Atkins Diet administration
  1. Carbohydrates intake will be restricted to 10 grams/ day. (Carbohydrate values of various food items will be explained in detail, and exchange lists provided. Four 2.5 grams carbohydrate exchange items will be allowed in a day.)
  2. Fats (e.g. cream, butter, oils, ghee) encouraged.
  3. Proteins (cheese, fish, eggs, chicken, soya products) unrestricted.
  4. Clear carbohydrate-fluids not restricted.
  5. Calcium and multivitamin supplementation will be provided.
  Other Names: Dietary intervention
  Arms: 1

SUMMARY:
Seizures are a frequent cause of morbidity in the pediatric age group. Uncontrolled seizures pose a variety of risks to children, including higher rates of mortality, developmental delay and/or regression, and cognitive impairment. The ketogenic diet is a well known treatment option for refractory epilepsy. However it is very restrictive and requires strict weighing of foods. The modified Atkins diet is a dietary therapy for intractable childhood epilepsy that was designed to be a less restrictive alternative to the traditional ketogenic diet. Early studies have demonstrated efficacy and safety.There are no randomized trials evaluating the efficacy of the modified Atkins diet in children with refractory epilepsy. Hence this study has been planned to investigate whether there are clear benefits in terms of seizure control in children with refractory epilepsy who are treated with the modified Atkins diet, versus controls.

DETAILED DESCRIPTION:
Several severe catastrophic epilepsies present in childhood, including severe infantile myoclonic epilepsy, Lennox Gastaut syndrome and myoclonic-astatic epilepsy (Doose syndrome). Seizures in these disorders are difficult to control; sometimes only at the expense of multiple and toxic levels of antiepileptic medications.Epilepsy surgery is feasible only in a very small number, also the costs are prohibitively high.

Uncontrolled seizures pose a variety of risks to children, including higher rates of mortality, developmental delay and/or regression, and cognitive impairment. Thus effective treatment to control seizures is fundamental to improving overall outcome in childhood epilepsy. The shortcomings of antiepileptic drug therapy and epilepsy surgery have made the need for alternative treatments.

The ketogenic diet is one of the oldest available treatments for epilepsy. It is a medically supervised high fat, low carbohydrate, and restricted protein diet that maintains a chronic state of ketosis while providing proteins and calories for adequate growth. The ketogenic diet compares favourably with the newer antiepileptic drugs (AED's) which have been developed for the treatment epilepsy in children Studies on the newer antiepileptic drugs such as vigabatrin, lamotrigine, tiagabine and gabapentin indicate that only 3% to 10% of all intractable patients achieve complete relief of seizures with the introduction of these newer drugs. Whereas with the ketogenic diet, 33% of patients with intractable epilepsy have more than 50% reduction in seizures and 15-20% become seizure free.Also, many of the children who are maintained on the diet are able to have their antiepileptic drugs decreased or withdrawn. This leads to improvement in alertness, behaviour and cognition.

The traditional ketogenic diet, with 4:1 ratio of fat: carbohydrate + protein has its drawbacks. It restricts calories and fluids, and requires weighing of foods. Protein is generally restricted to 1 g/kg/day, with the majority of remaining calories in the form of fat. This may lead to hypoproteinemia and growth problems. Hospitalization is generally advocated for diet initiation, both for fasting and non-fasting initiation. Side effects of the diet include kidney stones, constipation, acidosis, diminished growth, weight loss, and hyperlipidemia.

The modified Atkins diet is a nonpharmacologic therapy for intractable childhood epilepsy that was designed to be a less restrictive alternative to the traditional ketogenic diet. This diet is started on an outpatient basis without a fast, allows unlimited protein and fat, and does not restrict calories or fluids. Early studies have demonstrated efficacy and safety.13-20 However these studies have been uncontrolled, and have enrolled small numbers of patients. There are no randomized control trials evaluating the efficacy of the modified Atkins diet in children and adults with refractory epilepsy. Hence this study has been was planned to investigate whether there are clear benefits in terms of seizure control in children with refractory epilepsy who are treated with the modified Atkins diet, versus controls.

Eligible children will be randomized using computer generated random number tables in two groups: the intervention and the control arm. Both groups will undergo a baseline 4-week observation period, during which parents will be asked to maintain a daily seizure activity log; recording seizure type, duration and frequency. In the intervention arm, the children will start the modified Atkins diet after this 4-week baseline period. The control group will receive their normal diet with no dietetic input, and remain on the same on-going antiepileptic medication for the 3 months. Anti-epileptic medications will remain unchanged during the 3 month trial period in both groups, unless the change in AED regimen is medically indicated; e.g. drug side effects or status epilepticus; in which case standard therapy will be provided.

Children will be reviewed as outpatients at 1, 2 and 3 months. Urinary ketones will be checked at each hospital visit. A 3-day dietary intake chart will be reviewed at each visit to compute calorie and carbohydrate intake, and reinforce compliance. Weight will be checked at each visit.

Seizure frequencies will be recorded daily for the 4-week baseline period and the 3 month study period. At the end of the 3 month study period, the number of seizures in the preceding 28 days will be used to calculate the mean seizure number, which will be expressed as a percentage of the mean baseline number of daily seizures (ie, the number of seizures during the 4 weeks before the child started either the diet or the control phase of the study).No changes will be made to the child's antiepileptic medication during the 4-week baseline or the 3-month study periods, unless medically indicated; e.g. drug side effects, or status epilepticus; in which case standard therapy will be provided.

Tolerability of the diet and its side effects will be evaluated by means of parental interview at each visit: vomiting, lethargy, poor appetite, refusal to feed and constipation. Any other parental concerns or parental reports of side effects will also be noted.

ELIGIBILITY:
Inclusion Criteria:

* Seizures persisting daily or more than 7 per week despite the appropriate use of at least 3 anti-epileptic drugs.

Exclusion Criteria:

* Known or suspected inborn error of metabolism
* Clinical suspicion of metabolic disorder as evidenced by 2 or more of the following:

  * a history of parental consanguinity
  * prior affected siblings
  * unexplained vomiting
  * intermittent worsening of symptoms
  * recurrent episodes of lethargy
  * altered sensorium, or ataxia
  * hepatosplenomegaly on examination
* And/ or 2 or more of the following biochemical abnormalities

  * High blood ammonia (>80mmol/L)
  * High arterial lactate (>2 mmol/L)
  * metabolic acidosis (pH <7.2)
  * hypoglycaemia (blood sugar <40 mg/dl)
  * abnormal urinary aminoacidogram
  * presence of reducing sugars or ketones in urine
  * positive results on urine neurometabolic screening tests
* Motivational or psychosocial issues in the family which would preclude compliance
* Systemic illness- chronic hepatic, renal or pulmonary disease

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Reduction in seizure frequency at 3 months in the two groups: the modified Atkins diet group, and the control group. | 3 months

SECONDARY OUTCOMES:
Tolerability and the adverse effects of the modified Atkins diet. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Suvasini Sharma, MD, Principal Investigator — All India Institute of Medical Sciences; Sheffali Gulati, MD, Study Director — All India Institute of Medical Sciences; Anuja Agarwala, MSc, Study Chair — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Martin-McGill KJ, Bresnahan R, Levy RG, Cooper PN. Ketogenic diets for drug-resistant epilepsy. Cochrane Database Syst Rev. 2020 Jun 24;6(6):CD001903. doi: 10.1002/14651858.CD001903.pub5. PMID 32588435
- [Derived] Sharma S, Sankhyan N, Gulati S, Agarwala A. Use of the modified Atkins diet for treatment of refractory childhood epilepsy: a randomized controlled trial. Epilepsia. 2013 Mar;54(3):481-6. doi: 10.1111/epi.12069. Epub 2013 Jan 7. PMID 23294191